CLINICAL TRIAL: NCT00780962
Title: N-Acetylcysteine to Prevent Radiocontrast Nephropathy in Emergency Department Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Cumberland Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Nathan Shapiro, Associate Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2007P000095
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Results first posted 2018-01-31 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Radiocontrast Nephropathy
Keywords: NAC; Radiocontrast Nephropathy; N-Acetylcysteine; RCN; RCIN; Creatinine; Computerized Tomography; CT; Emergency Department; ED
MeSH Terms: conditions — Emergencies | interventions — Acetylcysteine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive either of two interventions: N-acetylcysteine (Treatment group) or Normal Saline (Placebo group).
  Patients in the treatment group will receive 3 g of Nacetylcysteine in 500mL normal saline (0.9% Sodium Chloride) solution during 30 minutes before contrast administration. After contrast administration, patients will receive a continuous infusion of 200mg of N-acetylcysteine per hour, administered as an infusion of 67 mL per hour of a solution of 3 g of N-acetylcysteine diluted to a total volume of 1,000 mL with normal saline solution.
  Patients in the placebo group will receive 500 mL of normal saline solution during 30 minutes before contrast administration and a continuous infusion of 67 mL per hour of normal saline solution after contrast administration.
  Patients in both arms will receive the postcontrast infusion (N-acetylcysteine or saline solution) for a minimum of 2 hours.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study medication (or placebo) will come premixed from the pharmacy. There will be no external marks on the medication (or placebo) that suggests its identity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N-Acetylcysteine group (Experimental): Subjects in this group will receive 3 grams of N-acetylcysteine in 500 cc normal saline (0.9% Sodium Chloride) over 30 minutes prior to contrast administration. After contrast administration, they will receive a continuous infusion of 200 mg N-acetylcysteine per hour. This dose will be administered as an infusion of 67 cc per hour of a solution of 3 grams of N-acetylcysteine in 1000 cc of normal saline. The infusion will be administered for a minimum of two hours and then stopped after 24 hours, or when the patient is discharged from the Emergency Department or the hospital, whichever comes first.
  Interventions: Drug: N-Acetylcysteine (NAC)
- 0.9% Sodium-chloride group (Placebo Comparator): Subjects in this group will receive 500 cc Normal Saline (0.9% Sodium Chloride) over 30 minutes prior to contrast administration. After contrast administration, they will receive a continuous infusion of 67 cc per hour of normal saline. The infusion will be administered for a minimum of two hours and then stopped after 24 hours, or when the patient is discharged from the Emergency Department or the hospital, whichever comes first.
  Interventions: Drug: 0.9% Sodium-chloride

INTERVENTIONS:
Drug: N-Acetylcysteine (NAC) — Experimental:
  * Before CT: 3 g NAC IV in 500 cc of 0.9% Sodium-chloride
  * After CT: 200 mg NAC/hour in 0.9% Sodium-chloride at 67 cc/hour for up to 24 hours.
  Other Names: Acetadote
  Arms: N-Acetylcysteine group
Drug: 0.9% Sodium-chloride — Placebo:
  * Before CT: 500 cc 0.9% Sodium-chloride
  * After CT: NS at 67 cc/hour for up to 24 hours.
  Other Names: Normal Saline
  Arms: 0.9% Sodium-chloride group

SUMMARY:
Multiple agents have been studied to prevent radiocontrast nephropathy. One of these agents is N-Acetylcysteine. Previous trials to assess N-Acetylcysteine's efficacy in the prevention of contrast nephropathy have been promising. However, previous studies have limited applicability to the Emergency Department (ED) patient population for two reasons:

* 1) Many of the pretreatment strategies employed in these studies take several hours or even days to perform, which is not feasible in acutely ill ED patients.
* 2) Most of these studies were conducted in patients undergoing cardiac catheterization. This may be a very different population than patients in the ED undergoing abdominal or chest computed tomography.

The investigators wish to study the efficacy of N-acetylcysteine as an agent to prevent radiocontrast nephropathy in ED patients undergoing computerized tomography. The investigators propose a randomized, double-blind, controlled trial comparing saline hydration plus N-acetylcysteine versus saline hydration alone. The hypothesis of this study is that N-acetylcysteine with normal saline will be more effective than saline alone in the prevention of radiocontrast nephropathy.

DETAILED DESCRIPTION:
Out of the approximately 110 million Emergency Department (ED) visits in the United States each year approximately 8.8 million people undergo Contrast-Enhanced Computerized Tomography (CT) studies in United States EDs each year (based on the investigators experience).

Radiocontrast nephropathy is a serious potential consequence associated with significant morbidity and mortality. Preliminary data suggests that the rate of Radiocontrast Induced Nephropathy after Emergency Department CT is approximately 5-7%. This figure, coupled with our estimate of 8.8 million contrast-enhanced CT studies, suggests that there are somewhere between 440,000 and 616,000 cases of radiocontrast nephropathy in the US each year that are caused by ED studies.

Multiple agents have been studied to prevent radiocontrast nephropathy. One of these agents is N-Acetylcysteine. There is inconclusive evidence about the benefit of this intervention. Some studies have shown that N-Acetylcysteine administered in either a high-dose intravenous protocol or a low-dose intravenous plus oral protocol may reduce the incidence of radiocontrast nephropathy in patients undergoing emergent cardiac catheterization, although other studies have found no benefit.

It is not clear, however, if these studies generalize to the ED patient undergoing emergency CT. ED patients often have different comorbidities or higher acuity which may limit the applicability in the ED patient population for two reasons:

* 1) Many of the pretreatment strategies employed in these studies take several hours or even days to perform, which is not feasible in acutely ill ED patients.
* 2) Most of these studies were conducted in patients undergoing cardiac catheterization. This may be a very different population than patients in the ED undergoing abdominal or chest computed tomography.

The investigators wish to study the efficacy of N-acetylcysteine as an agent to prevent radiocontrast nephropathy in ED patients undergoing computerized tomography. The investigators propose a randomized, double-blind, controlled trial comparing saline hydration plus N-acetylcysteine versus saline hydration alone. The hypothesis of this study is that N-acetylcysteine with normal saline will be more effective than saline alone in the prevention of radiocontrast nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a CT with intravenous contrast as part of clinical care
* 18 years of age or older
* Willingness to have a serum creatinine measured 48-72 hours after study
* Presence of one or more risk factors for radiocontrast nephropathy:

  * Creatinine greater than or equal to 1.4 mg/dL
  * Estimated Glomerular Filtration Rate (eGFR) of less than 60 mL/min/1.73m2
  * Diabetes Mellitus
  * Hypertension being treated with anti-hypertensive mediations
  * Coronary artery disease
  * Concurrent use of any of the following nephrotoxic drugs:

    * Cyclosporine A
    * Aminoglycosides
    * Amphotericin
    * Cisplatin
    * Non-steroidal anti-inflammatory drugs
    * Congestive heart failure (active or by history)
    * Older age (65 years of age or older)
    * Anemia (hematocrit < 30%)

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* End-stage renal disease currently undergoing regular hemodialysis
* Pregnant
* Known allergy to N-acetylcysteine
* Too unstable to wait for infusion of medication or placebo
* Treating physician using N-Acetylcysteine as part of clinical care

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2007-10-16 (Actual); Primary Completion 2010-08-09 (Actual); Study Completion 2010-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Traub, MD, Principal Investigator — Beth Israel Deaconess Medical Center, Boston
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baker CS, Wragg A, Kumar S, De Palma R, Baker LR, Knight CJ. A rapid protocol for the prevention of contrast-induced renal dysfunction: the RAPPID study. J Am Coll Cardiol. 2003 Jun 18;41(12):2114-8. doi: 10.1016/s0735-1097(03)00487-x. PMID 12821233
- [Background] Gupta R, Gurm HS, Bhatt DL, Chew DP, Ellis SG. Renal failure after percutaneous coronary intervention is associated with high mortality. Catheter Cardiovasc Interv. 2005 Apr;64(4):442-8. doi: 10.1002/ccd.20316. PMID 15789398
- [Background] Hipp A, Desai S, Lopez C, Sinert R. The incidence of contrast-induced nephropathy in trauma patients. Eur J Emerg Med. 2008 Jun;15(3):134-9. doi: 10.1097/MEJ.0b013e328270367d. PMID 18460952
- [Background] Kao LW, Kirk MA, Furbee RB, Mehta NH, Skinner JR, Brizendine EJ. What is the rate of adverse events after oral N-acetylcysteine administered by the intravenous route to patients with suspected acetaminophen poisoning? Ann Emerg Med. 2003 Dec;42(6):741-50. doi: 10.1016/s0196-0644(03)00508-0. PMID 14634597
- [Background] Kay J, Chow WH, Chan TM, Lo SK, Kwok OH, Yip A, Fan K, Lee CH, Lam WF. Acetylcysteine for prevention of acute deterioration of renal function following elective coronary angiography and intervention: a randomized controlled trial. JAMA. 2003 Feb 5;289(5):553-8. doi: 10.1001/jama.289.5.553. PMID 12578487
- [Background] Marenzi G, Assanelli E, Marana I, Lauri G, Campodonico J, Grazi M, De Metrio M, Galli S, Fabbiocchi F, Montorsi P, Veglia F, Bartorelli AL. N-acetylcysteine and contrast-induced nephropathy in primary angioplasty. N Engl J Med. 2006 Jun 29;354(26):2773-82. doi: 10.1056/NEJMoa054209. PMID 16807414
- [Background] Marenzi G, Lauri G, Assanelli E, Campodonico J, De Metrio M, Marana I, Grazi M, Veglia F, Bartorelli AL. Contrast-induced nephropathy in patients undergoing primary angioplasty for acute myocardial infarction. J Am Coll Cardiol. 2004 Nov 2;44(9):1780-5. doi: 10.1016/j.jacc.2004.07.043. PMID 15519007
- [Background] Merten GJ, Burgess WP, Gray LV, Holleman JH, Roush TS, Kowalchuk GJ, Bersin RM, Van Moore A, Simonton CA 3rd, Rittase RA, Norton HJ, Kennedy TP. Prevention of contrast-induced nephropathy with sodium bicarbonate: a randomized controlled trial. JAMA. 2004 May 19;291(19):2328-34. doi: 10.1001/jama.291.19.2328. PMID 15150204
- [Background] Rashid ST, Salman M, Myint F, Baker DM, Agarwal S, Sweny P, Hamilton G. Prevention of contrast-induced nephropathy in vascular patients undergoing angiography: a randomized controlled trial of intravenous N-acetylcysteine. J Vasc Surg. 2004 Dec;40(6):1136-41. doi: 10.1016/j.jvs.2004.09.026. PMID 15622367
- [Background] Rihal CS, Textor SC, Grill DE, Berger PB, Ting HH, Best PJ, Singh M, Bell MR, Barsness GW, Mathew V, Garratt KN, Holmes DR Jr. Incidence and prognostic importance of acute renal failure after percutaneous coronary intervention. Circulation. 2002 May 14;105(19):2259-64. doi: 10.1161/01.cir.0000016043.87291.33. PMID 12010907
- [Background] Smilkstein MJ, Bronstein AC, Linden C, Augenstein WL, Kulig KW, Rumack BH. Acetaminophen overdose: a 48-hour intravenous N-acetylcysteine treatment protocol. Ann Emerg Med. 1991 Oct;20(10):1058-63. doi: 10.1016/s0196-0644(05)81352-6. PMID 1928874
- [Result] Traub SJ, Mitchell AM, Jones AE, Tang A, O'Connor J, Nelson T, Kellum J, Shapiro NI. N-acetylcysteine plus intravenous fluids versus intravenous fluids alone to prevent contrast-induced nephropathy in emergency computed tomography. Ann Emerg Med. 2013 Nov;62(5):511-520.e25. doi: 10.1016/j.annemergmed.2013.04.012. Epub 2013 Jun 14. PMID 23769807
- [Result] Traub SJ, Kellum JA, Tang A, Cataldo L, Kancharla A, Shapiro NI. Risk factors for radiocontrast nephropathy after emergency department contrast-enhanced computerized tomography. Acad Emerg Med. 2013 Jan;20(1):40-5. doi: 10.1111/acem.12059. PMID 23570477

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6,977 patients of 2 Emergency Departments at 2 tertiary care, urban university hospitals (Beth Israel Deaconess Medical Center in Boston, MA and Carolinas Medical Center in Charlotte, NC) were assessed for Eligibility between October 2007 and August 2010.
Groups:
- N-Acetycysteine Group: Participants in this group received 3 grams of N-acetylcysteine in 500 cc Normal Saline (0.9% Sodium Chloride) over 30 minutes prior to contrast administration. After contrast administration, participants received a continuous infusion of 200 mg N-acetylcysteine per hour, administered as an infusion of 67 cc per hour of a solution of 3 grams of N-acetylcysteine diluted in a total volume of 1000 cc of normal saline.
- 0.9% Sodium-chloride Group: Patients in the placebo group received 500 mL of normal saline solution during 30 minutes before contrast administration and a continuous infusion of 67 mL per hour of normal saline solution after contrast administration
Period: Overall Study
Arm/Group | N-Acetycysteine Group | 0.9% Sodium-chloride Group
Started | 200 | 199
Second Blood Draw (Outcome Measurement) | 185 | 172
Completed | 185 | 172
Not Completed | 15 | 27

BASELINE CHARACTERISTICS:
Population: 399 subjects were consented to participate in the study, of whom 357 (89.4%) completed a second blood draw to determine outcome and were included in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | N-Acetycysteine Group | 0.9% Sodium-chloride Group | Total
Number analyzed (Participants) | 200 | 199 | 399
Age, Continuous [Mean (Full Range); unit: years] | 61.5 [28 to 95] | 59.7 [18 to 94] | 60.6 [18 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 113 | 237
  Male | 76 | 86 | 162
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 199 | 199 | 398
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 50 | 47 | 97
  White | 138 | 142 | 280
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 8 | 19
Baseline Creatinine [Mean (Full Range); unit: mg/dL] — Population: 399 subjects were enrolled in the study, of whom 357 (89.4%) completed a second blood draw. Reported here the Baseline Creatinine serum level (first value meassured) of the participants who completed the second blood draw.
  mg/dL
    number analyzed (Participants) | 185 | 172 | 357
    (all) | 1.0 [0.5 to 1.9] | 0.99 [0.5 to 1.8] | 0.99 [0.5 to 1.9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Contrast-induced Nephropathy
Description: Contrast-induced nephropathy was defined as an increase in serum creatinine level of greater than or equal to 0.5 mg/dL or an increase of 25% above baseline. The primary outcome was measured by the change in serum creatinine level from the pre-radiocontrast baseline to the serum creatinine level measured 48 to 72 hours after radiocontrast administration.
Time Frame: 48-72 hours
Population: Out of 399 subjects who consented to participate in the study, only 357 (89.4%) had a second blood creatinine levels measurement done between 48 to 72h.
Measure: Count of Participants; unit: Participants
Arm/Group | N-Acetycysteine Group | 0.9% Sodium-chloride Group
Number analyzed (Participants) | 185 | 172
Participants | 14 | 12
Statistical Analysis 1: Comparison: N-Acetycysteine Group vs 0.9% Sodium-chloride Group; The study was powered to find a 10% absolute risk reduction in the rate of contrast-induced nephropathy (a=.05, 90% power). We initially estimated the need for 600 patients and repowered to 800 patients after the 1st interim analysis. The study was halted for futility at the 2nd interim analysis. Reported here 357 (89.4%) of the 399 enrolled subjects who completed a second blood draw at the time the study closed; Test type: Superiority; p > 0.5, Wald; Percentage Difference = 0.6, 95% CI 2-sided [-4.8 to 6.0]

ADVERSE EVENTS:
Time Frame: Study participants were monitored during the infusions. Also, we performed a follow-up telephone call to identify patients who had clinically significant renal injury beyond the 72-hour period.
Description: Participants were closely monitored by the clinical team. Infusions were discontinued in the event of symptomatic hypotension requiring treatment, altered mental status, respiratory distress, pulmonary edema, oropharyngeal edema or bronchospasm requiring treatment, severe urticaria or patient discomfort, or any other event considered severe enough by the clinical team treating the patient to require discontinuation.
Arm/Group | N-Acetycysteine Group | 0.9% Sodium-chloride Group
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/199
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/199
Other Adverse Events (participants affected / at risk) | 13/200 | 17/199
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetycysteine Group (N=200) | 0.9% Sodium-chloride Group (N=199)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Flushing (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Other (General disorders) | 3 (3) | 4 (4)

LIMITATIONS AND CAVEATS:
Our results were obtained in patients considered to be at relatively low risk for contrast-induced nephropathy and should not be extended to patients who might be at higher risk for it.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No